CLINICAL TRIAL: NCT07386977
Title: Influence of Visual Feedback on Angular Error in Knee Joint Position Sense
Brief Title: Effects of Visual Feedback on Angular Error
Status: Active, not recruiting | Type: Observational
Sponsor: Lokman Hekim University (Other Government)
Responsible Party: Principal Investigator, Seda BAKTIR, Assist. Prof., Lokman Hekim University
Other Study IDs: LHU-FTR-ZSBD-04
Record Dates: First submitted 2026-01-28; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Knee Osteoarthritis; Gonarthrosis
Keywords: knee osteoarthritis; proprioception; angular error; joint position sense; gonarthrosis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1-Knee Joint Position Evaluation with Visual Input: The participant was instructed, in a seated position, to extend the knee from the starting position of 90° knee flexion until reaching the target angle of 30° knee flexion.
- 2-Knee Joint Position Evaluation without Visual Input: The participant was instructed, in a prone position, to move the knee from the starting position of 90° knee flexion to the target angle of 30° knee flexion.

SUMMARY:
With this study is to evaluate knee joint position sense in patients with gonarthrosis under conditions with and without visual input.

DETAILED DESCRIPTION:
Knee injuries, such as ligament ruptures or cartilage damage, can significantly impair proprioception. Previous studies have shown that individuals with knee injuries often exhibit reduced proprioceptive acuity, which may lead to altered movement patterns and consequently increase the risk of re-injury. Moreover, even asymptomatic knees may demonstrate proprioceptive errors due to underlying, undiagnosed conditions such as osteoarthritis, suggesting that proprioceptive dysfunction itself may contribute to injury occurrence.

The role of visual input in the assessment of proprioception is also of considerable importance. Studies have demonstrated that visual feedback can enhance proprioceptive accuracy by providing additional sensory information that supports joint position sense. In contrast, the absence of visual cues has been associated with increased joint positioning errors, indicating that proprioception is not solely dependent on proprioceptive feedback but is also influenced by visual input. Investigating the interaction between visual and proprioceptive information is therefore crucial for the effective regulation of motor control.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 80 years,
* A confirmed diagnosis of knee osteoarthritis,
* Absence of any health condition that could interfere with the measurement procedures.

Exclusion Criteria:

* Refusal to participate in the study,
* Presence of a diagnosed neurological disorder that could affect the measurements,
* Presence of cardiopulmonary instability that could influence the measurements,
* History of knee-related trauma within the past year,
* Receipt of physiotherapy or rehabilitation treatment within the past year,
* History of knee-related surgery,
* Inability to follow verbal instructions due to insufficient cognitive function.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with knee osteoarthritis according to Kellgren-Lawrence grades 1-3 were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Proprioception Measurement | Each measurement was repeated three times with 1-minute intervals between trials. A 2-minute rest period was allowed between conditions involving changes in visual input.
  During the measurement, the inclinometer was aligned so that its axis passed through the knee joint line, and it was positioned on the proximal one-third of the fibula and secured in place using a strap. Measurements were performed both with visual input and with visual input eliminated. After reaching the target position, the participant maintained the final position for 5 seconds before returning to the starting position.

CONTACTS AND LOCATIONS:
Overall Officials: ZAHİDE SEDA BAKTIR DOĞAN, Assist. Prof, Principal Investigator — Lokman Hekim University
Locations (1):
- Lokman Hekim University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We are planning not to share this data not to declare the data of our participants with any third group.